CLINICAL TRIAL: NCT03971695
Title: Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Doses of BI 706321 in Healthy Male Subjects (Single-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study to Test How Well Healthy Men Tolerate Different Doses of BI 706321
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1425-0001; 2019-000888-25 (EudraCT Number)
Record Dates: First submitted 2019-05-31; First posted 2019-06-03 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Part I - Placebo oral solution (Placebo Comparator): Part I - Placebo oral solution matching BI 706321 as single dose taken orally with 240 milliliter (mL) of water after an overnight fast of at least 10 hours. Placebo subjects were randomised in a 3:1 ratio over the matching BI 706321 arms.
  Interventions: Drug: Placebo
- Part I - 0.3 mg BI 706321 oral solution (Experimental): Part I - 1.2 mL oral solution of 0.25 mg/mL (0.3 milligram (mg) BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours
  Interventions: Drug: BI 706321
- Part I - 0.6 mg BI 706321 oral solution (Experimental): Part I - 2.4 mL oral solution of 0.25 mg/mL (0.6 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 706321
- Part I - 1.2 mg BI 706321 oral solution (Experimental): Part I - 4.8 mL oral solution of 0.25 mg/mL (1.2 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 706321
- Part I - Placebo capsules (Placebo Comparator): Part I - Placebo capsules BI 706321 as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours. Placebo subjects were randomised in a 3:1 ratio over the matching BI 706321 arms.
  Interventions: Drug: Placebo
- Part I - 2 mg BI 706321 capsules (Experimental): Part I - 2 capsules of 1 mg (2 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 706321
- Part I - 4 mg BI 706321 capsules (Experimental): Part I - 4 capsules of 1 mg (4 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 706321
- Part I - 8 mg BI 706321 capsules (Experimental): Part I - 8 capsules of 1 mg (8 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 706321
- Part I - 15 mg BI 706321 capsules (Experimental): Part I - 3 capsules of 5 mg (15 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 706321
- Part I - 25 mg BI 706321 capsules (Experimental): Part I - 5 capsules of 5 mg (25 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 706321
- Part II - Test 1 (T1), fasted, tablets (Experimental): Part II - Test 1 (T1), fasted: 2 tablets of 2 mg (4 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours
  Interventions: Drug: BI 706321
- Part II - Test 2 (T2), fed, tablets (Experimental): Part II - Test 2 (T2), fed: 2 tablets of 2 mg (4 mg BI 706321) as single dose taken orally with 240 mL of water after a high-fat, high-calorie breakfast.
  Interventions: Drug: BI 706321
- Part II - Reference (R), fasted, capsules (Experimental): Part II - Reference (R), fasted: 4 capsules of 1 mg (4 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours.
  Interventions: Drug: BI 706321

INTERVENTIONS:
Drug: BI 706321 — Capsule or Oral Solution
  Arms: Part I - 0.3 mg BI 706321 oral solution; Part I - 0.6 mg BI 706321 oral solution; Part I - 1.2 mg BI 706321 oral solution; Part I - 15 mg BI 706321 capsules; Part I - 2 mg BI 706321 capsules; Part I - 25 mg BI 706321 capsules; Part I - 4 mg BI 706321 capsules; Part I - 8 mg BI 706321 capsules; Part II - Reference (R), fasted, capsules; Part II - Test 1 (T1), fasted, tablets; Part II - Test 2 (T2), fed, tablets
Drug: Placebo — Capsule or Oral solution
  Arms: Part I - Placebo capsules; Part I - Placebo oral solution

SUMMARY:
The main objectives are:

* Part I: To investigate safety, tolerability, and pharmacokinetics (PK) of BI 706321 in healthy male subjects following oral administration of single rising doses.
* Part II: The relative bioavailability of BI 706321 after administration of tablets and capsules under fasted conditions will be compared with each other and the effect of food on the tablet bioavailability will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (BP, PR, oral body temperature), 12-lead ECG, and clinical laboratory tests
* Age of 18 to 45 years (inclusive) in Part I and of 18 to 55 years (inclusive) in Part II
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with GCP and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), (PR), oral body temperature or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 24 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male subjects with WOCBP partner who are unwilling to use male contraception (condom or sexual abstinence) from time point of administration of trial medication until 30 days thereafter. Sperm donation is not allowed from the time point of drug administration until 30 days thereafter.
* ALT (alanine transaminase), AST (aspartate transaminase), or creatinine exceed upper limit of normal range at screening, confirmed by a repeat test
* During COVID-19 pandemic: laboratory test indicative of an ongoing SARS-CoV-2 infection

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2020-12-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Part I of the trial was designed as randomised, placebo-controlled, and single-blind, within parallel dose groups.
  Part II of the trial was designed as a randomised, open-label, 3-way crossover to compare the treatments T1 and R (comparison A) and T2 and T1 (comparison B).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Part II - R-T1-T2: Part II - R-T1-T2 - Reference (R), fasted: 4 capsules of 1 mg (4 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours. Test 1 (T1), fasted: 2 tablets of 2 mg (4 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours. Test 2 (T2), fed: 2 tablets of 2 mg (4 mg BI 706321) as single dose taken orally with 240 mL of water after a high-fat, high-calorie breakfast. Treatments in Part II were separated by a washout period of at least 12 days.
- Part II - T1-T2-R: Part II - T1-T2-R - Test 1 (T1), fasted: 2 tablets of 2 mg (4 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours. Test 2 (T2), fed: 2 tablets of 2 mg (4 mg BI 706321) as single dose taken orally with 240 mL of water after a high-fat, high-calorie breakfast. Reference (R), fasted: 4 capsules of 1 mg (4 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours. Treatments in Part II were separated by a washout period of at least 12 days.
- Part II - T2-R-T1: Part II - T2-R-T1 - Test 2 (T2), fed: 2 tablets of 2 mg (4 mg BI 706321) as single dose taken orally with 240 mL of water after a high-fat, high-calorie breakfast. Reference (R), fasted: 4 capsules of 1 mg (4 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours. Test 1 (T1), fasted: 2 tablets of 2 mg (4 mg BI 706321) as single dose taken orally with 240 mL of water after an overnight fast of at least 10 hours. Treatments in Part II were separated by a washout period of at least 12 days.
Period: Part I and Period 1 of Part II
Arm/Group | Part I - Placebo Oral Solution | Part I - 0.3 mg BI 706321 Oral Solution | Part I - 0.6 mg BI 706321 Oral Solution | Part I - 1.2 mg BI 706321 Oral Solution | Part I - Placebo Capsules | Part I - 2 mg BI 706321 Capsules | Part I - 4 mg BI 706321 Capsules | Part I - 8 mg BI 706321 Capsules | Part I - 15 mg BI 706321 Capsules | Part I - 25 mg BI 706321 Capsules | Part II - R-T1-T2 | Part II - T1-T2-R | Part II - T2-R-T1
Started | 6 | 6 | 6 | 5 | 9 | 6 | 6 | 6 | 5 | 6 | 4 | 4 | 4
Completed | 6 | 6 | 6 | 5 | 9 | 6 | 6 | 6 | 5 | 6 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: End of Part I and Part II - Washout
Arm/Group | Part I - Placebo Oral Solution | Part I - 0.3 mg BI 706321 Oral Solution | Part I - 0.6 mg BI 706321 Oral Solution | Part I - 1.2 mg BI 706321 Oral Solution | Part I - Placebo Capsules | Part I - 2 mg BI 706321 Capsules | Part I - 4 mg BI 706321 Capsules | Part I - 8 mg BI 706321 Capsules | Part I - 15 mg BI 706321 Capsules | Part I - 25 mg BI 706321 Capsules | Part II - R-T1-T2 | Part II - T1-T2-R | Part II - T2-R-T1
Started | 6 | 6 | 6 | 5 | 9 | 6 | 6 | 6 | 5 | 6 | 4 | 4 | 4
Completed | 0 (Participants did not take part in the crossover part (Part II) of the study.) | 0 (Participants did not take part in the crossover part (Part II) of the study.) | 0 (Participants did not take part in the crossover part (Part II) of the study.) | 0 (Participants did not take part in the crossover part (Part II) of the study.) | 0 (Participants did not take part in the crossover part (Part II) of the study.) | 0 (Participants did not take part in the crossover part (Part II) of the study.) | 0 (Participants did not take part in the crossover part (Part II) of the study.) | 0 (Participants did not take part in the crossover part (Part II) of the study.) | 0 (Participants did not take part in the crossover part (Part II) of the study.) | 0 (Participants did not take part in the crossover part (Part II) of the study.) | 4 | 4 | 4
Not Completed | 6 | 6 | 6 | 5 | 9 | 6 | 6 | 6 | 5 | 6 | 0 | 0 | 0
Not completed — Did not participate in part II of study | 6 | 6 | 6 | 5 | 9 | 6 | 6 | 6 | 5 | 6 | 0 | 0 | 0
Period: Part II - Period 2
Arm/Group | Part I - Placebo Oral Solution | Part I - 0.3 mg BI 706321 Oral Solution | Part I - 0.6 mg BI 706321 Oral Solution | Part I - 1.2 mg BI 706321 Oral Solution | Part I - Placebo Capsules | Part I - 2 mg BI 706321 Capsules | Part I - 4 mg BI 706321 Capsules | Part I - 8 mg BI 706321 Capsules | Part I - 15 mg BI 706321 Capsules | Part I - 25 mg BI 706321 Capsules | Part II - R-T1-T2 | Part II - T1-T2-R | Part II - T2-R-T1
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II - Washout (of at Least 12 Days)
Arm/Group | Part I - Placebo Oral Solution | Part I - 0.3 mg BI 706321 Oral Solution | Part I - 0.6 mg BI 706321 Oral Solution | Part I - 1.2 mg BI 706321 Oral Solution | Part I - Placebo Capsules | Part I - 2 mg BI 706321 Capsules | Part I - 4 mg BI 706321 Capsules | Part I - 8 mg BI 706321 Capsules | Part I - 15 mg BI 706321 Capsules | Part I - 25 mg BI 706321 Capsules | Part II - R-T1-T2 | Part II - T1-T2-R | Part II - T2-R-T1
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II - Period 3
Arm/Group | Part I - Placebo Oral Solution | Part I - 0.3 mg BI 706321 Oral Solution | Part I - 0.6 mg BI 706321 Oral Solution | Part I - 1.2 mg BI 706321 Oral Solution | Part I - Placebo Capsules | Part I - 2 mg BI 706321 Capsules | Part I - 4 mg BI 706321 Capsules | Part I - 8 mg BI 706321 Capsules | Part I - 15 mg BI 706321 Capsules | Part I - 25 mg BI 706321 Capsules | Part II - R-T1-T2 | Part II - T1-T2-R | Part II - T2-R-T1
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug. The treatment assignment was determined based on the first treatment the subjects received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part I - Placebo Oral Solution | Part I - 0.3 mg BI 706321 Oral Solution | Part I - 0.6 mg BI 706321 Oral Solution | Part I - 1.2 mg BI 706321 Oral Solution | Part I - Placebo Capsules | Part I - 2 mg BI 706321 Capsules | Part I - 4 mg BI 706321 Capsules | Part I - 8 mg BI 706321 Capsules | Part I - 15 mg BI 706321 Capsules | Part I - 25 mg BI 706321 Capsules | Part II - R-T1-T2 | Part II - T1-T2-R | Part II - T2-R-T1 | Total
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 9 | 6 | 6 | 6 | 5 | 6 | 4 | 4 | 4 | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (4.7) | 28.8 (4.8) | 30.3 (3.9) | 32.8 (4.4) | 32.3 (5.9) | 29.2 (4.9) | 35.3 (6.8) | 30.2 (6.2) | 29.6 (2.9) | 32.2 (7.8) | 39.8 (6.4) | 42.0 (11.5) | 35.0 (12.5) | 32.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 5 | 9 | 6 | 6 | 6 | 5 | 6 | 4 | 4 | 4 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 6 | 5 | 9 | 6 | 6 | 6 | 5 | 6 | 4 | 4 | 4 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 5 | 9 | 6 | 6 | 6 | 5 | 6 | 4 | 4 | 4 | 73
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Part I: Percentage of Subjects With Drug-related Adverse Events
Description: Part I: Percentage of subjects with drug-related adverse events.
Time Frame: Between intake of trial medication and the individual subject's end of trial, up to 22 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Part I - Placebo Oral Solution | Part I - 0.3 mg BI 706321 Oral Solution | Part I - 0.6 mg BI 706321 Oral Solution | Part I - 1.2 mg BI 706321 Oral Solution | Part I - Placebo Capsules | Part I - 2 mg BI 706321 Capsules | Part I - 4 mg BI 706321 Capsules | Part I - 8 mg BI 706321 Capsules | Part I - 15 mg BI 706321 Capsules | Part I - 25 mg BI 706321 Capsules
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 9 | 6 | 6 | 6 | 5 | 6
Percentage of participants | 16.7 | 16.7 | 0.0 | 0.0 | 11.1 | 0.0 | 0.0 | 16.7 | 20.0 | 33.3

2. Primary Outcome: Part II: Area Under the Concentration-time Curve of BI 706321 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz)
Description: Part II: Area under the concentration-time curve of BI 706321 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz).
Time Frame: Within 3 hours before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 34, 48, 72, 168 hours after drug administration.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set included all subjects in the TS who provided at least 1 PK endpoint that was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomol/liter
Arm/Group | Part II - Test 1 (T1), Fasted, Tablets | Part II - Test 2 (T2), Fed, Tablets | Part II - Reference (R), Fasted, Capsules
Number analyzed (Participants) | 12 | 12 | 12
hour*nanomol/liter | 150 (27.5) | 138 (29.9) | 150 (29.5)
Statistical Analysis 1: Comparison: Part II - Test 1 (T1), Fasted, Tablets vs Part II - Reference (R), Fasted, Capsules; Analysis of variance (ANOVA) on the logarithmic scale including effects for 'sequence', 'subjects nested within sequences', 'period', and 'treatment'. Confidence intervals were calculated based on the residual error from the ANOVA; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 100.26, 90% CI 2-sided [90.18 to 111.48] — Intra-individual geometric coefficient of variance (gCV) = 14.2. Ratio is T1/R
Statistical Analysis 2: Comparison: Part II - Test 1 (T1), Fasted, Tablets vs Part II - Test 2 (T2), Fed, Tablets; [analysis description as in outcome 2, analysis 1]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 91.63, 90% CI 2-sided [85.37 to 98.35] — Intra-individual geometric coefficient of variance (gCV) = 9.5. Ratio is T2/T1

3. Primary Outcome: Part II: Maximum Measured Concentration of BI 706321 in Plasma (Cmax)
Description: Part II: Maximum measured concentration of BI 706321 in plasma (Cmax).
Time Frame: Within 3 hours before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 34, 48, 72, 168 hours after drug administration.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/liter
Arm/Group | Part II - Test 1 (T1), Fasted, Tablets | Part II - Test 2 (T2), Fed, Tablets | Part II - Reference (R), Fasted, Capsules
Number analyzed (Participants) | 12 | 12 | 12
nanomol/liter | 5.90 (47.8) | 4.57 (33.6) | 6.02 (41.1)
Statistical Analysis 1: Comparison: Part II - Test 1 (T1), Fasted, Tablets vs Part II - Reference (R), Fasted, Capsules; [analysis description as in outcome 2, analysis 1]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 98.01, 90% CI 2-sided [84.20 to 114.08] — Intra-individual geometric coefficient of variance (gCV) = 20.5. Ratio is T1/R
Statistical Analysis 2: Comparison: Part II - Test 1 (T1), Fasted, Tablets vs Part II - Test 2 (T2), Fed, Tablets; [analysis description as in outcome 2, analysis 1]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 77.52, 90% CI 2-sided [68.11 to 88.22] — Intra-individual geometric coefficient of variance (gCV) = 17.4. Ratio is T2/T1

4. Secondary Outcome: Part I: Area Under the Concentration-time Curve of BI 706321 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Part I: Area under the concentration-time curve of BI 706321 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: Within 3 hours before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 34, 48, 168 hours after drug administration.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomol/liter
Arm/Group | Part I - 0.3 mg BI 706321 Oral Solution | Part I - 0.6 mg BI 706321 Oral Solution | Part I - 1.2 mg BI 706321 Oral Solution | Part I - 2 mg BI 706321 Capsules | Part I - 4 mg BI 706321 Capsules | Part I - 8 mg BI 706321 Capsules | Part I - 15 mg BI 706321 Capsules | Part I - 25 mg BI 706321 Capsules
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 5 | 6 | 5 | 6
hour*nanomol/liter | NA (NA) — Not calculated due to insufficient concentration data above the lower limit of assay quantitation | NA (NA) — Not calculated due to insufficient concentration data above the lower limit of assay quantitation | NA (NA) — Not calculated due to insufficient concentration data above the lower limit of assay quantitation | NA (NA) — Not calculated due to insufficient concentration data above the lower limit of assay quantitation | 151 (33.1) | 314 (25.7) | 618 (36.1) | 1130 (24.2)

5. Secondary Outcome: Part I: Maximum Measured Concentration of BI 706321 in Plasma (Cmax)
Description: Part I: Maximum measured concentration of BI 706321 in plasma (Cmax).
Time Frame: Within 3 hours before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 34, 48, 168 hours after drug administration.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomol/liter
Arm/Group | Part I - 0.3 mg BI 706321 Oral Solution | Part I - 0.6 mg BI 706321 Oral Solution | Part I - 1.2 mg BI 706321 Oral Solution | Part I - 2 mg BI 706321 Capsules | Part I - 4 mg BI 706321 Capsules | Part I - 8 mg BI 706321 Capsules | Part I - 15 mg BI 706321 Capsules | Part I - 25 mg BI 706321 Capsules
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 5 | 6 | 5 | 6
nanomol/liter | 0.388 (32.8) | 0.781 (21.4) | 1.02 (40.0) | 2.27 (30.1) | 5.19 (38.6) | 11.8 (41.6) | 24.6 (43.0) | 41.1 (32.1)

6. Secondary Outcome: Part I: Time From Dosing to the Maximum Measured Concentration of BI 706321 in Plasma (Tmax)
Description: Part I: Time from dosing to the maximum measured concentration of BI 706321 in plasma (tmax).
Time Frame: Within 3 hours before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 34, 48, 168 hours after drug administration.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part I - 0.3 mg BI 706321 Oral Solution | Part I - 0.6 mg BI 706321 Oral Solution | Part I - 1.2 mg BI 706321 Oral Solution | Part I - 2 mg BI 706321 Capsules | Part I - 4 mg BI 706321 Capsules | Part I - 8 mg BI 706321 Capsules | Part I - 15 mg BI 706321 Capsules | Part I - 25 mg BI 706321 Capsules
Number analyzed (Participants) | 6 | 6 | 5 | 6 | 5 | 6 | 5 | 6
hours | 5.61 (16.7) | 5.25 (51.6) | 5.22 (31.8) | 5.24 (51.6) | 4.91 (22.3) | 4.12 (43.7) | 3.37 (70.7) | 3.64 (62.1)

7. Secondary Outcome: Part II: Area Under the Concentration-time Curve of BI 706321 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Part II: Area under the concentration-time curve of BI 706321 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
Time Frame: Within 3 hours before and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 34, 48, 72, 168 hours after drug administration.
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanomol/liter
Arm/Group | Part II - Test 1 (T1), Fasted, Tablets | Part II - Test 2 (T2), Fed, Tablets | Part II - Reference (R), Fasted, Capsules
Number analyzed (Participants) | 12 | 12 | 12
hour*nanomol/liter | 169 (26.1) | 154 (28.0) | 171 (27.7)
Statistical Analysis 1: Comparison: Part II - Test 1 (T1), Fasted, Tablets vs Part II - Reference (R), Fasted, Capsules; [analysis description as in outcome 2, analysis 1]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 96.42, 90% CI 2-sided [86.96 to 106.90] — Intra-individual geometric coefficient of variance (gCV) = 13.9. Ratio is T1/R
Statistical Analysis 2: Comparison: Part II - Test 1 (T1), Fasted, Tablets vs Part II - Test 2 (T2), Fed, Tablets; [analysis description as in outcome 2, analysis 1]; Test type: Other; Adjusted geometric mean (gMean) ratio(%) = 91.27, 90% CI 2-sided [85.40 to 97.54] — Intra-individual geometric coefficient of variance (gCV) = 8.9. Ratio is T2/T1

ADVERSE EVENTS:
Time Frame: Between (first) intake of trial medication and the time of the next administration of trial medication (Part II) or the individual subject's end of trial (Part I and Part II). Up to 22 days.
Description: Treated set (TS): The TS included all subjects who were randomised and treated with at least 1 dose of trial drug. The treatment assignment was determined based on the first treatment the subjects received.
Groups:
- Placebo Total: All subjects treated with placebo oral solution or placebo capsules groups.
- BI 706321 Total Part I: All subjects in Part I treated with BI 706321.
- Total Part I: All subjects in Part I.
- BI 706321 Total Part II: All subjects in Part II treated with BI 706321.
- BI 706321 Total: All subjects in Part I and II treated with BI 706321.
- Total: All subjects in Part I and II.
Arm/Group | Part I - Placebo Oral Solution | Part I - Placebo Capsules | Part I - 0.3 mg BI 706321 Oral Solution | Part I - 0.6 mg BI 706321 Oral Solution | Part I - 1.2 mg BI 706321 Oral Solution | Part I - 2 mg BI 706321 Capsules | Part I - 4 mg BI 706321 Capsules | Part I - 8 mg BI 706321 Capsules | Part I - 15 mg BI 706321 Capsules | Part I - 25 mg BI 706321 Capsules | Part II - Test 1 (T1), Fasted, Tablets | Part II - Test 2 (T2), Fed, Tablets | Part II - Reference (R), Fasted, Capsules | Placebo Total | BI 706321 Total Part I | Total Part I | BI 706321 Total Part II | BI 706321 Total | Total
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/12 | 0/12 | 0/12 | 0/15 | 0/46 | 0/61 | 0/12 | 0/58 | 0/73
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 0/6 | 0/6 | 0/5 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/12 | 0/12 | 0/12 | 0/15 | 0/46 | 0/61 | 0/12 | 0/58 | 0/73
Other Adverse Events (participants affected / at risk) | 3/6 | 3/9 | 3/6 | 2/6 | 1/5 | 0/6 | 3/6 | 1/6 | 3/5 | 2/6 | 1/12 | 2/12 | 2/12 | 6/15 | 15/46 | 21/61 | 4/12 | 19/58 | 25/73
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part I - Placebo Oral Solution (N=6) | Part I - Placebo Capsules (N=9) | Part I - 0.3 mg BI 706321 Oral Solution (N=6) | Part I - 0.6 mg BI 706321 Oral Solution (N=6) | Part I - 1.2 mg BI 706321 Oral Solution (N=5) | Part I - 2 mg BI 706321 Capsules (N=6) | Part I - 4 mg BI 706321 Capsules (N=6) | Part I - 8 mg BI 706321 Capsules (N=6) | Part I - 15 mg BI 706321 Capsules (N=5) | Part I - 25 mg BI 706321 Capsules (N=6) | Part II - Test 1 (T1), Fasted, Tablets (N=12) | Part II - Test 2 (T2), Fed, Tablets (N=12) | Part II - Reference (R), Fasted, Capsules (N=12) | Placebo Total (N=15) | BI 706321 Total Part I (N=46) | Total Part I (N=61) | BI 706321 Total Part II (N=12) | BI 706321 Total (N=58) | Total (N=73)
Photokeratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 3 | 3
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Pre-existing condition improved (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Puncture site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 2
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Scar (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Myosclerosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 3
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/95/NCT03971695/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT03971695/SAP_001.pdf